CLINICAL TRIAL: NCT02938767
Title: Carotid Intima-media Thickness and Coronary Flow Reserve as Cardiovascular Event and Mortality Predictors in Peritoneal Dialysis Patients: Results of Seven-year Follow-up From a Single Center
Brief Title: Carotid Intima-media Thickness as Cardiovascular Mortality Predictor in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, MD Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University
Other Study IDs: 3221
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Myocardial Infarction
Keywords: peritoneal dialysis; carotid intima-media thickness; coronary flow reserve; cardiovascular mortality
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hemogram, serum creatinine, uric asid, calcium, phosphorus and albumin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- peritoneal dialysis patients: 37 peritoneal dialysis patients followed at the Istanbul Medical Faculty from October 1994 to October 2011
- renal transplant recipients: 20 renal transplant recipients followed at the Istanbul Medical Faculty from October 1994 to October 2011 setted as the control group

SUMMARY:
Cardiovascular (CV) disease is the main cause of death in patients on dialysis. The aim of this study is the long-term prognostic values of carotid intima-media thickness and coronary flow reserve in cardiovascular mortality of peritoneal dialysis patients.

DETAILED DESCRIPTION:
Endothelial dysfunction (ED) is a precursor and cause of cardiovascular diseases. Defining of endothelial thickness and coronary microvascular function could be useful for detecting ED. Endothelial dysfunction could be assessed by coronary flow reserve (CFR), carotid intima media thickness (IMT). Repeating measurement of IMT and CFR could be predictor of cardiovascular events and mortality in peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients whose followed up at least six months from October 1994 to October 2011 (for study group)
* Kidney transplant recipients whose followed up at least six months from October 1994 to October 2011 (for control group)

Exclusion Criteria:

* diabetes mellitus
* valvular heart disease,
* any prior coronary intervention and congestive heart failure
* Patients whose left anterior descending coronary artery (LAD) could not be visualized adequately by Doppler echocardiography were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were treated by peritoneal dialysis or followed up as kidney transplant recipient at the Istanbul Medical Faculty from October 1994 to October 2011. Two groups were established for trial as peritoneal dialysis patients and renal transplant recipients. Patients had follow up shorter than six months and missing data not included in the trial
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diseases morbidity | 10-15 years

SECONDARY OUTCOMES:
Patient Survival | 10-15 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No